CLINICAL TRIAL: NCT02512926
Title: Phase I Study of Carfilzomib in Combination With Cyclophosphamide and Etoposide for Children With Relapsed and Refractory Solid Tumors and Leukemias
Brief Title: Carfilzomib in Combination With Cyclophosphamide and Etoposide for Children
Acronym: POE14-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Pediatric Oncology Experimental Therapeutics Investigators' Consortium (Unknown); Amgen (Industry)
Responsible Party: Principal Investigator, Norman J. Lacayo, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-37313; PEDSVAR0042 (Other: Stanford - OnCore); NCT03273829 (obsolete NCT alias)
Record Dates: First submitted 2015-07-21; First posted 2015-07-31 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Relapsed Solid Tumors; Refractory Solid Tumors; Relapsed Leukemia; Refractory Leukemia
Keywords: Solid Tumors; Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Leukemia; Recurrence | interventions — carfilzomib; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib in combination with cyclophosphamide and etoposide
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib in combination with cyclophosphamide and etoposide for children with relapsed and refractory solid tumors and leukemias
Drug: Cyclophosphamide
Drug: Etoposide

SUMMARY:
This study evaluates the use of carfilzomib in combination with cyclophosphamide and etoposide for children with relapsed/refractory solid tumors or leukemia. The medications cyclophosphamide and etoposide are standard drugs often used together for the treatment of cancer in children with solid tumors or leukemia.

Carfilzomib is FDA (Food and Drug Administration) approved in the United States for adults with multiple myeloma (a type of cancer). However, this drug is not approved to treat children with relapsed/refractory solid tumors or leukemia. With this research, we plan to determine the DLTs and MTD of Carfilzomib given in combination with cyclophosphamide and etoposide in pediatric patients with relapsed/refractory leukemias and solid tumors.

DETAILED DESCRIPTION:
Part 1 of the study will include a dose escalation based on Dose limiting toxicities (DLTs) until the MTD or highest dose level is reached, whichever comes first.

At the MTD or highest dose level (if no MTD is reached), an additional 6 patients will be enrolled to further evaluate safety of the regimen (Part 2).

Part 2 of this study will enroll additional patients at the highest tolerable dose found in Part 1 in order to get more information on side effects and make sure the dose is tolerable

Once an MTD is determined for Strata A or B, if the Study Principal Investigator determines that the study treatment should not be further pursued due to safety or enrollment barriers, the expansion Part or the study will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have either of the following:

   1. Relapsed/refractory leukemia in 2nd or greater relapse or who have failed at least one re-induction attempt after relapse or for refractory disease. Patients must meet the WHO classification with ≥ 5% blasts in the bone marrow or must have definitive extramedullary disease (e.g. chloromas, skin lesions). Patients may have asymptomatic CNS 1 or CNS 2 disease, but not CNS 3 or symptomatic CNS disease.

      OR
   2. Relapsed/refractory non-CNS solid tumor that has not responded or has relapsed and for which no standard treatment is available. Patients may not have primary CNS tumors or CNS metastases. Lymphoma patients are permitted. Patients do not need to have measurable disease.
2. Age 6 months - 29.99 years at enrollment
3. Life expectancy ≥ 3 months
4. Lansky or Karnofsky ≥50
5. Prior therapy

   1. Patient must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, radiotherapy, or surgery prior to study entry.
   2. Myelosuppressive therapy- At least 14 days must have elapsed since the administration of previous therapy. Six weeks must have elapsed from the administration of nitrosureas or mitomycin C. For patients with ALL on maintenance therapy, they may be eligible if 7 days have elapsed and they are recovered from the toxic effects of the chemotherapy. This restriction does not include intrathecal chemotherapy, which is permitted.
   3. Biologic agents- At least 14 days must have elapsed since the completion of therapy with a biologic agent such as a monoclonal antibody. Seven days must have elapsed since the last dose of retinoids
   4. Radiation therapy - At least 14 days must have elapsed for local XRT. At least 90 days must have elapsed if prior radiation to ≥50% of the pelvis, the spine, or other substantial bone marrow radiation including TBI.
   5. Hematopoietic growth factors- At least 7 days must have elapsed since the last dose of G-CSF or GM-CSF. At least 14 days must have elapsed since last dose of pegfilgrastim (Neulasta®).
6. Patient must be ≥ 3 months from hematopoietic stem cell transplant, must not have active GVHD, and must be off all immunosuppression
7. Organ function:

   1. Either a serum creatinine ≤ ULN for age, or calculated or measured GFR ≥ 70 mL/min/1.73 m2
   2. Total bilirubin ≤ 1.5 x ULN for age, direct bilirubin ≤ ULN for age
   3. AST and ALT ≤ 3 x ULN for age unless elevation can be clearly attributed to liver leukemia or metastases
   4. ECHO shortening fraction ≥ 27%
   5. Pulse Oximetry measurement ≥ 95% saturation without supplemental oxygen
8. Bone marrow function:

   1. Hgb ≥10 g/dL - can be transfused
   2. Plts ≥ 75,000 - cannot be transfused (must be ≥ 7 days from last plt transfusion)
   3. ANC ≥ 750 - cannot be transfused (must be ≥ 72 hours from last neutrophil infusion)

   However, the plt and ANC requirements can be waived if low counts thought to be secondary to leukemia or tumor bone marrow infiltration
9. Reproductive function:

   1. Female patients of childbearing potential must have a negative serum pregnancy test confirmed within 7 days prior to enrollment
   2. Female patients with infants must agree not to breastfeed their infants while on the study
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 3 months after study treatment
10. Written informed consent

Exclusion Criteria:

1. Prior treatment with carfilzomib
2. Known allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
3. Down syndrome
4. Fanconi Anemia or other underlying bone marrow failure syndrome
5. Pregnant or lactating females
6. Known history of Hepatitis B or C or HIV
7. Patient with any significant concurrent illness
8. Patient with uncontrolled systemic fungal, bacterial, viral or other infection with ongoing signs/symptoms despite appropriate treatment
9. Patient with illness, psychiatric disorder or social issue that could compromise patient safety or compliance with the protocol treatment or procedures, or interfere with the consent, study participation, follow-up, or interpretation of study results.

Ages: 6 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
To determine the DLTs and MTD of carfilzomib given in combination with cyclophosphamide and etoposide in pediatric patients with relapsed/refractory leukemias and solid tumors | 30 Days post treatment initiation

SECONDARY OUTCOMES:
To evaluate toxicities of carfilzomib in the pediatric population when combined with conventional chemotherapy. | Treatment initiation through 30 days post treatment
  Record AEs and SAEs
Determine patient response rate (CR, PR, SD, PD) with this regimen | Treatment initiation through 30 days post treatment
To measure if circulating plasma proteosome (cProt) levels post treatment correlate with response to therapy and overall survival. | Treatment initiation through 30 days post treatment
To measure if the levels of proteasome activity and resistance to carfilzomib correlates with toxicity and/or response to treatment | Treatment initiation through 30 days post treatment
To measure if inhibition of proteasome activity by carfilzomib results in alteration in a number of autophagy and apoptosis related proteins, providing means to evaluate correlates of activity of carfilzomib | Treatment initiation through 30 days post treatment
To measure the level of proteosome inhibition in patient PBMCs before and during treatment by determination of the level of protein ubiquitination | Treatment initiation through 30 days post treatment
To determine in vitro sensitivity of patient leukemias and solid tumors to carfilzomib alone and in combination with study chemotherapeutic agents in order to generate a predictive model of drug sensitivity | Treatment initiation through 30 days post treatment
To perform whole exome sequencing (WES) and RNA seq on patient leukemia and solid tumor samples and WES on germ line DNA in order to determine potential mechanisms of drug sensitivity or resistance | Treatment initiation through 30 days post treatment

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University School of Medicine and Stanford Cancer Institute, Palo Alto, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Boklan J, Langevin AM, Bielamowicz K, Neville K, Trippett T, Brown V, DuBois SG, Eshun F, Gelfond J, Zomet A, Narendran A, Lacayo NJ. A Phase I Study of Carfilzomib with Cyclophosphamide and Etoposide in Relapsed and Refractory Leukemia and Solid Tumors. Cancers (Basel). 2025 Sep 6;17(17):2924. doi: 10.3390/cancers17172924. PMID 40941020
- See also: Cancers 2025, 17(17), 2924 — https://pubmed.ncbi.nlm.nih.gov/40941020/